CLINICAL TRIAL: NCT01086982
Title: Pharmacodynamics Of Product Octreotide Acetate Lar 30 Mg, Imported And Distributed By The Laboratory Chemical Pharm. Bergamo, Compared To Product Sandostatin LAR®30 MG Manufactured By Novartis Biosciences S/A
Brief Title: Pharmacodynamics Of Product Octreotide Acetate Lar 30 Mg Compared To Product Sandostatin LAR ®
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OCTBER0409; Version 3 (Other: Protocol Version)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

ARMS (2):
- Octreotide acetate LAR 30 MG (Experimental): Test
  Interventions: Drug: Octreotide acetate LAR
- Sandostatin LAR ® (octreotide acetate LAR) 30 MG (Active Comparator)
  Interventions: Drug: Sandostatin LAR ® (octreotide acetate LAR) 30 MG

INTERVENTIONS:
Drug: Octreotide acetate LAR — 30 mg, single dose
  Arms: Octreotide acetate LAR 30 MG
Drug: Sandostatin LAR ® (octreotide acetate LAR) 30 MG — 30 mg, single dose
  Arms: Sandostatin LAR ® (octreotide acetate LAR) 30 MG

SUMMARY:
Check the pharmacodynamics of the drug octreotide acetate LAR 30 mg imported and distributed by Chemical Laboratory Pharmaceutical Bergamo Ltda. compared to the drug Sandostatin LAR ® (octreotide acetate 30 mg) manufactured by Novartis Biociências S / A, using as activity analysis of growth hormone (GH) and growth factor insulin-like 1 (IGF-1 ) after a single dose of the drug in patients with acromegaly

DETAILED DESCRIPTION:
Secondly, it will be observed safety (tolerability) in clinical patients by comparing the clinical and laboratory parameters before and after the study and the incidence of adverse events after a single dose

ELIGIBILITY:
Inclusion Criteria:

- Accept the Terms of Consent;

* be aged over 18, regardless of sex;
* Patients with acromegaly who presented GH levels ≥ 2.5 ng / mL or no suppression of GH levels to less than 1 ng / mL after tolerance test glucose and IGF-I levels for age and sex;
* Patients undergoing hypophysectomy followed by radiotherapy or not and to keep níves increased GH and IGF-I;
* Patients waiting hypophysectomy with increased levels of GH and IGF-I

Exclusion Criteria:

* Have participated in any experimental study or have ingested any drug trial within six months prior to the start of the study;
* Have made use of medications that influence the results, regular 4 weeks prior to the start of the study or having used any medication a week before the start of the study;
* Have been treated with somastostatina analog or dopamine agonist in the last 2 months;
* Present history of myocardial infarction, angina and / or heart failure;
* Patients who present calculation of the gallbladder and have not undergone cholecystectomy;
* Pregnant women and nursing;
* Patients who have allergies to medicine;
* Patients with a history of acute pancreatitis;
* Patient with altered levels of amylase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05

PRIMARY OUTCOMES:
Quantification of serum levels of GH and IGF-I. | Before drug administration, after drug administration, 1, 3, 7, 14, 21, 28, 35, 42, 49, 56 and 63 days after.

SECONDARY OUTCOMES:
Occurrence and severity of side effects during use of the product in order to ensure the security of it. | After drug administration, 1, 3, 7, 14, 21, 28, 35, 42, 49, 56 and 63 days after.

CONTACTS AND LOCATIONS:
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil